CLINICAL TRIAL: NCT06983587
Title: Study to Establish Reference Curves for Bone Mineral Density (BMD) and Body Composition (BC) in Women Aged 20-89 MONIKA
Brief Title: Reference Curves for Bone Mineral Density and Body Composition in Women Aged 20-89
Acronym: MONIKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other); Hôpital Edouard Herriot (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IDIL/2023/VB-01
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Bone Density
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Women aged 20-29 (Other): This group will be used to construct the T-score equation, and thus define the thresholds for osteopenia and osteoporosis. To ensure adequate precision for this T-score, 175 subjects will be included in this age group. With this number of subjects, the following accuracies for two of the sites of interest (hip and L1-L4) are expected:
  For the hip, the expected bone mineral density value is 0.95 (SD=0.11) according to local data consistent with Arlot et al. Inclusion of 175 subjects would give a ½ width 95% confidence interval (IC95%) of the mean would be around 0.016, and the half width standard deviation of 0.012 For L1-L4, the expected bone mineral density value is 0.99 (SD=0.11) according to local data consistent with Arlot et al. The ½ width of the 95% confidence interval (IC95%) of the mean would be around 0.016, and the half-width standard deviation of 0.012.
  Interventions: Radiation: Bone densitometry scan
- Women aged 30-39 (Other): For the 30-39 age group, only 25 subjects will be included, given the constancy of bone mineral density in this age group compared with the 20-29 age group. In addition, the results of the analyses will take the form of a Z-score equation, estimated using a regression method (i.e. overall and not a z-score per age group). As there will be many subjects under 30 and over 40, this will ensure (by interpolation) an equivalent precision in these age brackets to that of the adjacent age categories.
  Interventions: Radiation: Bone densitometry scan
- Women aged 40-49 (Other): Group including 50 subjects.
  Interventions: Radiation: Bone densitometry scan
- Women aged 50-59 (Other): Group including 50 subjects.
  Interventions: Radiation: Bone densitometry scan
- Women aged 60-69 (Other): Group including 50 subjects.
  Interventions: Radiation: Bone densitometry scan
- Women aged 70-79 (Other): Group including 50 subjects.
  Interventions: Radiation: Bone densitometry scan
- Women aged 80-89 (Other): Only 25 subjects will be included in this age group for reasons of feasibility.
  Interventions: Radiation: Bone densitometry scan

INTERVENTIONS:
Radiation: Bone densitometry scan — Each study participant will undergo a bone density measurement scan. The equipment used in this study will be the STRATOS DR X-ray bone densitometer (APELEM, 9 Avenue du Canal Philippe Lamour, 30660 Gallargues-le-Montueux, France). This device is indicated for diagnosing osteoporosis, assessing the risk of fracture in weakened bone areas, monitoring bone density, monitoring body composition and diagnosing vertebral anomalies (vertebral compression, fractures).
  In general, the time for a scan is less than 1 min for the spine, less than than 1 min for the femur, less than 1 min for the forearm and around 4 min for the whole body.
  The total duration of the patient's participation in this research will be approximately 2 hours.
  Other Names: Dual-energy X-ray absorptiometry (DEXA or DXA)

SUMMARY:
Up-to-date normalcy curves for bone mineral density and body composition (fat and lean mass), are currently lacking. DMS IMAGING is therefore financing the MONIKA study, with Nîmes University Hospital as sponsor.

Some 425 healthy female volunteers aged 20 to 89 will be recruited from three centers (Nîmes, Montpellier and Lyon). A bone density scan at various bone sites (femur, rachis, radius and whole body) will provide up-to-date normalcy curves for bone mineral density as well as body composition (fat and lean mass). These measurements should help to better understand bone physiology and the links that may exist between bone tissue and muscle and adipose tissue.

This is a prospective multicenter cross-sectional descriptive study of healthy female volunteers. The study population is made up of healthy female volunteers from Europe, the Middle East and North Africa aged between 20 and 89, stratified into 7 age groups.

DETAILED DESCRIPTION:
Bone densitometry using dual-photon X-ray absorptiometry (DXA) is the standard technique for measuring bone mineral density. According to the International Osteoporosis Foundation (IOF), if a single site is to be preferred, it should be the total hip or femoral neck, using a single NHANES III reference curve. It should be stressed, however, that this curve was obtained from a North American population with anthropometric parameters, notably body mass index (BMI), that differ from those of European populations, and more particularly of European, Middle Eastern and North African origin.

So far, only one reference curve has been obtained in France, from the OFELY study in 1993.

Given the age of this cohort and the possibility of changes in BMI over time in the population of European, Middle Eastern and North African origin, but even more so, the impossibility of transposing this curve onto new DXAs of different brands, new reference curves need to be developed. DMS IMAGING is therefore financing the MONIKA study, with Nîmes University Hospital as sponsor.

As part of this study, some 425 healthy female volunteers aged between 20 and 89 will be recruited from three centers (Nîmes, Montpellier, Lyon). A DXA examination at various bone sites (femur, rachis, radius and whole body) will provide up-to-date normalcy curves for BMD, but also for body composition (fat and lean mass), which are currently lacking. Access to this population could also enable us to better understand bone physiology and the links that may exist between bone tissue and muscle and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic origin European, Middle Eastern, North African and whose 2 parents are from Europe, Middle East, North Africa only as there is a difference in BMD according to ethnicity
* Person affiliated to or benefiting from a social security scheme
* Free, informed consent signed by the participant and the investigator (on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients presenting one of the following major risk factors:
* Fragility fracture defined as a spontaneous or low-kinetic fracture (≤ one fall from height)
* Hip fracture in a first-degree relative
* Early menopause (< age 40), Hysterectomy (complete < age 40), Primary amenorrhea (absence of menstruation before age 15), Current amenorrhea of more than 3 months without contraceptive if patient is under age 40
* Treatments : Prolonged corticosteroid therapy > 3 months or > 1 g (cumulative dose)
* Immobilization of more than 3 months, less than 12 months old
* Patients presenting one of the following pathologies affecting bone, muscle or adipose tissue:
* Chronic inflammatory bowel disease (IBD) (Crohn's disease, ulcerative colitis) and untreated celiac disease
* Renal insufficiency on dialysis or patients with nephrology follow-up
* Known hypercalciuria
* Osteomalacia, rickets, osteogenesis imperfecta
* Osteopathy (Paget's disease, osteopetrosis, etc.)
* Chronic inflammatory rheumatism
* Haemopathy, neoplasia
* Hepatic insufficiency or chronic hepatitis
* Endocrinopathy: dysthyroidism, hypogonadism, hypercorticism, untreated acromegaly.
* Anorexia nervosa
* Hyperparathyroidism (even if controlled)
* History of digestive surgery (bariatric, gastrectomy, digestive resection other than appendectomy, etc.)
* History of organ transplant
* Chronic infectious disease (HIV, etc.)
* Weight loss of more than 10 kg in the last 6 months
* Paresis, marked lameness or unloading of a limb or prolonged immobilisation of more than one month in the last 12 months

All patients on any treatment that may affect bone mass or body composition:

* Biphosphonates (Alendronate (Fosamax® and generics), Risedronate (Actonel® and generics), Zoledronate (Aclasta® and generics)
* Teriparatide (Forsteo®)
* Denosumab (Prolia®)
* Selective oestrogen receptor modulator (Clomifen, Tamoxifen, Toremifen, Raloxifen)
* Anabolic steroids.
* Strontium ranelate
* Carbamazepine
* Phenobarbital
* Immunosuppressants
* Antiepileptics

All patients with one of the following anomalies in the measurement area:

* Major deformities of the wrist, hip or vertebrae
* Compression of the vertebral bodies, cementoplasty
* Prosthesis, implant (breast, buttock, etc.), foreign body
* Hip paraosteoarthropathy
* Injection of radiological contrast product, barium enema, nuclear medicine examination within 10 days

Miscellaneous :

* Intensive sport (more than 10 h/week).
* Extreme BMI (BMI < 18, BMI > 35 kg/m²).
* Loss of autonomy
* Pregnant, parturient or breast-feeding woman
* Participation in an interventional study involving a drug or medical device or a category 1 RIPH in the 3 months prior to inclusion.

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — People with vaginas. Healthy female volunteers.
Enrollment: 425 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density of the femoral neck: Left side | Day 0, day of inclusion
  Bone mineral density (BMD in g/cm2) for the construction of Z score and T score
Bone mineral density of the femoral neck: Right side | Day 0, day of inclusion
  Bone mineral density (BMD in g/cm2) for the construction of Z score and T score
Bone mineral density of the femoral neck: Lumbar spine (L1 - L4) | Day 0, day of inclusion
  Bone mineral density (BMD in g/cm2) for the construction of Z score and T score
Bone mineral density of the femoral neck: Forearm | Day 0, day of inclusion
  Bone mineral density (BMD in g/cm2) for the construction of Z score and T score
Bone mineral density of the femoral neck: Whole body | Day 0, day of inclusion
  Bone mineral density (BMD in g/cm2) for the construction of Z score and T score

SECONDARY OUTCOMES:
Percentage body fat: left hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in %
Body fat: left hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Percentage body fat: right hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in %
Body fat: right hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Muscle mass: left hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Muscle mass: right hip | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Percentage body fat in the region of the lumbar spine (L1 - L4) | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in %
Body fat in the region of the lumbar spine (L1 - L4) | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Muscle mass in the region of the lumbar spine (L1 - L4) | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Percentage body fat: forearm | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in %
Body fat: forearm | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Muscle mass: forearm | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Percentage body fat: whole body | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in %
Body fat: whole body | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg
Muscle mass: whole body | Day 0, day of inclusion
  Measured automatically by the STRATOS DR X-ray bone densitometer in kg

OTHER OUTCOMES:
Weight of participants | Day 0, day of inclusion
  The weight of each participant will be recorded in kg
Height of participants | Day 0, day of inclusion
  The height of each participant will be recorded in cm
Body Mass Index of participants | Day 0, day of inclusion
  The body mass index (BMI) of each participant will be calculated as follows : BMI = weight [kg] / height 2 [m2]

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital, Montpellier, Hérault
  - Hôpital E Herriot UMR_S 1033, Lyon

IPD SHARING:
Plan to Share IPD: No
All data will be managed by the BESPIM (Biostatistics, Epidemiology, Public Health & Innovations in Methodology, Nîmes University Hospital). The conditions for the transfer of all or part of the research database are decided by the research sponsor and are the subject of a written contract.